CLINICAL TRIAL: NCT03305341
Title: Conducting an Initial Small, Controlled Clinical Pharmacology Trial to Assess for Therapeutic Biologics Activity (Proof-of-Concept) That Suggests the Potential for Clinical Benefits of COVID-19 Patients With Controlled Cancers.
Brief Title: Proof-of-Concept Clinical Pharmacology Trial for COVID-19 Antigen Presentation Therapeutic Biologic Mix
Acronym: COVSP-BCG
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IND165646; FWA00015357 (Registry Identifier: DHHS, OHRP); IRB00009424 (Registry Identifier: IRB, DHHS); IORG0007849 (Registry Identifier: IORG, DHHS); NPI-1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI-1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IND165646 (Registry Identifier: IND, FDA)
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Covid19
Keywords: Gene Mutation; Antigen Presentation; APC; Spike; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Intervention Model Description: Single Usage / Single Dosage
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assess for therapeutic biologics activity (proof-of-concept) (Experimental): Therapeutic Biological Product Mix activity - NOVAVAX COVID-19 VACCINE 1.0 mL add into BCG Organism 50 MG
  Interventions: Biological: COVID-19 Therapeutic Biologic Mix - NOVAVAX COVID-19 VACCINE plus BCG Vaccine Mix for percutaneous use

INTERVENTIONS:
Biological: COVID-19 Therapeutic Biologic Mix - NOVAVAX COVID-19 VACCINE plus BCG Vaccine Mix for percutaneous use — * By the percutaneous route with the multiple puncture device
  * NOVAVAX COVID-19 VACCINE 1.0 mL plus BCG Organism 50 MG Mix
  Other Names: NOVAVAX COVID-19 VACCINE plus BCG Vaccine Mix

SUMMARY:
Conducting an initial small, controlled clinical pharmacology trial to assess for therapeutic biologics activity (proof-of-concept) that suggests the potential for clinical benefit of COVID-19 patients with controlled cancers.

1. Treat Infection of Multiple Gene Mutation COVID-19 Virus Strains.
2. Activate Human Antigen Presentation Reaction to COVID-19 Specific Antigen.
3. The human antigen presenting cells (APCs) can take up and process COVID-19 target antigen protein into small peptide fragments, and then COVID-19 virus can be killed by APCs directly.

DETAILED DESCRIPTION:
* Conducting an initial small, controlled trial to assess therapeutic biologics activity (proof-of-concept) that suggests the potential for clinical benefit of COVID-19 patients with controlled cancers.
* 20 Moderate COVID-19 patients with controlled cancers
* Moderate COVID-19
* Positive testing by standard RT-PCR assay or equivalent testing
* Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion
* Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥ 20 breaths per minute, saturation of oxygen (SpO2) > 93% on room air at sea level, heart rate ≥ 90 beats per minute
* No clinical signs indicative of Severe or Critical Illness Severity
* Novavax COVID-19 Vaccine 1.0 mL plus BCG Organism 50 MG Mix
* By the percutaneous route with the multiple puncture device
* Negative testing COVID-19 by standard RT-PCR assay or equivalent testing after injection 3 weeks.
* Positive IGRA blood test with COVID-19 spike protein antigen after percutaneous use 21 days.
* Our trial duration will be 4 weeks.

ELIGIBILITY:
* Conducting an initial small, controlled trial to assess therapeutic biologics activity (proof-of-concept) that suggests the potential for clinical benefit of COVID-19 patients with controlled cancers.
* 20 Moderate COVID-19 patients with controlled cancers

Inclusion Criteria:

* Controlled Cancers
* Moderate COVID-19
* Positive testing by standard RT-PCR assay or equivalent testing
* Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion
* Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥ 20 breaths per minute, saturation of oxygen (SpO2) > 93% on room air at sea level, heart rate ≥ 90 beats per minute
* No clinical signs indicative of Severe or Critical Illness Severity

Exclusion Criteria:

* 1. Uncontrolled Cancers
* 2. Severe or Critical Illness Severity
* 3. Pregnancy
* 4. Breast-feeding
* 5. The patients with other serious inter-current illness
* 6. Serious Allergy
* 7. Serious Bleed Tendency
* 8. The prohibition of the biological product

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Moderate COVID-19: | Duration at least 28 days
  * 20 Moderate COVID-19 patients with controlled cancers
  * Moderate COVID-19
  * Positive testing by standard RT-PCR assay
  * Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion
  * Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥ 20 breaths per minute, saturation of oxygen (SpO2) > 93% on room air at sea level, heart rate ≥ 90 beats per minute
  * No clinical signs indicative of Severe or Critical Illness Severity
Rate of Positive COVID-19 nucleic acid: | Duration at least 28 days
  * 20 Moderate COVID-19 patients with controled cancers
  * Positive testing COVID-19 by standard RT-PCR assay immediately
  * COVID-19 nucleic acid testing, assessed by RT-PCR Assay Kit
  * Rate of Positive COVID-19 nucleic acid must be 100%
Rate of Negative COVID-19 nucleic acid | Duration at least 28 days
  * 20 Moderate COVID-19 patients with controlled cancers
  * NOVAVAX COVID-19 VACCINE 1.0 mL plus BCG Organism 50 MG Mix
  * By the percutaneous route with the multiple puncture device
  * Negative COVID-19 by standard RT-PCR assay after percutaneous use 3 weeks
  * COVID-19 nucleic acid testing, assessed by RT-PCR Assay Kit
  * Rate of Negative COVID-19 nucleic acid will be more than 80%
20 COVID-19 Participants with IGRA blood test with COVID-19 spike protein antigen | Duration at least 28 days
  Positive IGRA blood test with COVID-19 spike protein antigen after percutaneous use 21 days
20 COVID-19 Participants with IGRA blood test with TB antigens | Duration at least 28 days
  * Negative IGRA blood test with TB antigens before percutaneous use
  * Positive IGRA blood test with TB antigens after percutaneous use 21 days

CONTACTS AND LOCATIONS:
Overall Officials: HAN XU, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. (MIDI) - IORG0007849; HAN XU, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. (MIDI) - IORG0007849; HAN XU, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. (MIDI) - IORG0007849
Locations (1):
- Medicine Invention Design Incorporation (MIDI) - IORG0007849, North Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Netea MG, Dominguez-Andres J, Barreiro LB, Chavakis T, Divangahi M, Fuchs E, Joosten LAB, van der Meer JWM, Mhlanga MM, Mulder WJM, Riksen NP, Schlitzer A, Schultze JL, Stabell Benn C, Sun JC, Xavier RJ, Latz E. Defining trained immunity and its role in health and disease. Nat Rev Immunol. 2020 Jun;20(6):375-388. doi: 10.1038/s41577-020-0285-6. Epub 2020 Mar 4. PMID 32132681
- [Background] Sanchez-Ramon S, Conejero L, Netea MG, Sancho D, Palomares O, Subiza JL. Trained Immunity-Based Vaccines: A New Paradigm for the Development of Broad-Spectrum Anti-infectious Formulations. Front Immunol. 2018 Dec 17;9:2936. doi: 10.3389/fimmu.2018.02936. eCollection 2018. PMID 30619296
- [Background] Guevara-Hoyer K, Saz-Leal P, Diez-Rivero CM, Ochoa-Grullon J, Fernandez-Arquero M, Perez de Diego R, Sanchez-Ramon S. Trained Immunity Based-Vaccines as a Prophylactic Strategy in Common Variable Immunodeficiency. A Proof of Concept Study. Biomedicines. 2020 Jul 9;8(7):203. doi: 10.3390/biomedicines8070203. PMID 32660100
- [Background] Keech C, Albert G, Cho I, Robertson A, Reed P, Neal S, Plested JS, Zhu M, Cloney-Clark S, Zhou H, Smith G, Patel N, Frieman MB, Haupt RE, Logue J, McGrath M, Weston S, Piedra PA, Desai C, Callahan K, Lewis M, Price-Abbott P, Formica N, Shinde V, Fries L, Lickliter JD, Griffin P, Wilkinson B, Glenn GM. Phase 1-2 Trial of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine. N Engl J Med. 2020 Dec 10;383(24):2320-2332. doi: 10.1056/NEJMoa2026920. Epub 2020 Sep 2. PMID 32877576
- [Background] Wollina U. Challenges of COVID-19 pandemic for dermatology. Dermatol Ther. 2020 Sep;33(5):e13430. doi: 10.1111/dth.13430. Epub 2020 Apr 30. PMID 32314460
- [Background] Catala Gonzalo A, Galvan Casas C. COVID-19 and the Skin. Actas Dermosifiliogr (Engl Ed). 2020 Jul-Aug;111(6):447-449. doi: 10.1016/j.ad.2020.04.007. Epub 2020 May 13. No abstract available. English, Spanish. PMID 32401723
- [Background] Guarneri C, Rullo EV, Pavone P, Berretta M, Ceccarelli M, Natale A, Nunnari G. Silent COVID-19: what your skin can reveal. Lancet Infect Dis. 2021 Jan;21(1):24-25. doi: 10.1016/S1473-3099(20)30402-3. Epub 2020 May 18. No abstract available. PMID 32437697
- [Background] Freeman EE, McMahon DE, Lipoff JB, Rosenbach M, Kovarik C, Takeshita J, French LE, Thiers BH, Hruza GJ, Fox LP; American Academy of Dermatology Ad Hoc Task Force on COVID-19. Pernio-like skin lesions associated with COVID-19: A case series of 318 patients from 8 countries. J Am Acad Dermatol. 2020 Aug;83(2):486-492. doi: 10.1016/j.jaad.2020.05.109. Epub 2020 May 30. PMID 32479979
- See also: FWA00015357 — http://ohrp.cit.nih.gov/search
- See also: IRB00009424 — http://ohrp.cit.nih.gov/search
- See also: IORG0007849 — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03305341/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03305341/SAP_001.pdf
  • Informed Consent Form (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03305341/ICF_002.pdf